CLINICAL TRIAL: NCT03605147
Title: The Effect of Calcium β-hydroxy-β-methylbutyrate Supplementation in Sarcopenia in Liver Cirrhosis：A Randomized Double-blind Controlled Trial
Brief Title: The Effect of Calcium β-hydroxy-β-methylbutyrate (CaHMB) Supplementation in Sarcopenia in Liver Cirrhosis
Acronym: CaHMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIR-CAHMB-001
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Sarcopenia; Cirrhosis, Liver
Keywords: HMB; sarcopenia; liver cirrhosis; chronic liver disease; malnutrition; muscle wasting
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis; Malnutrition; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaHMB (Experimental): CaHMB Group (n=60) will receive CaHMB twice a day and a late evening snack every night for 12 weeks. A specialized, ready-to-drink liquid with 34 kcal, 8.5 g carbohydrate, 1.5g calcium-HMB. The late evening snack is a drink with low-Glycemic Index carbohydrate with 112 kcal.
  Interventions: Dietary Supplement: CaHMB
- Control (Active Comparator): Control Group (n=60) will receive placebo twice a day and placebo every night for 12 weeks with similar composition but without HMB. The late evening snack is a drink with low-Glycemic Index carbohydrate with 112 kcal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CaHMB — Supplements, labeled only with the identification number of the participant, will be provided to the participants in the Department of Gastroenterology of Zhongshan Hospital. After 4 weeks, subjects will receive medical center visit to evaluate the compliance and side effects. After 12 weeks, changes in body composition will be assessed by abdominal CT. An online application will be used to monitor the compliance everyday.Their diets will be recorded by a nutritionist. Blood will be collected pre- and post treatment. Extensive laboratory tests will be performed.
  Arms: CaHMB
Dietary Supplement: Placebo — Supplements, labeled only with the identification number of the participant, will be provided to the participants in the Department of Gastroenterology of Zhongshan Hospital. After 4 weeks, subjects will receive medical center visit to evaluate the compliance and side effects. After 12 weeks, changes in body composition will be assessed by CT. An online application will be used to monitor the compliance everyday.Their diets will be recorded by a nutritionist. Blood will be collected pre- and post treatment. Extensive laboratory tests will be performed.
  Arms: Control

SUMMARY:
This study is to evaluate the effect of CaHMB in the treatment of sarcopenia in liver cirrhosis.

DETAILED DESCRIPTION:
The study is a randomized double-blind controlled trial. Patients randomly enter into two treatment groups: 1) the CaHMB group and 2) the placebo group. Treatment allocation is by block randomization, with an one-to-one ratio for CaHMB and placebo. The results are concealed in opaque envelopes. Patients will report their daily diets with an online software. Patients will come for clinic after 4 weeks and 12 weeks, receiving laboratory tests and sarcopenia evaluation, and events of primary and secondary outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed of cirrhosis with imaging or liver biopsy;
2. diagnosis of portal hypertension with endoscopy or radiography；
3. assessed total muscle mass at the level of L3 (<42 cm2/m2 for male and <38 cm2/m2 for female)
4. has signed an informed consent form.

Exclusion Criteria:

1. diagnosed as hepatic cell cancer;
2. complicated with malignancy, renal failure, diabetes mellitus;
3. comorbidities including heart failure or pulmonary disease;
4. current use of drugs that affect skeletal muscle metabolism;
5. be allergic to the experimental food;
6. participated other clinical trials in the past 3 months;
7. other conditions that researchers consider not suitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Changes in skeletal muscle mass | Baseline and 12 weeks
  Changes of total muscle mass at the level of L3 in CT, analysed by the total cross-sectional area of muscle in centimetres squared (cm2)

SECONDARY OUTCOMES:
Changes in total body weight | Baseline and 12 weeks
  Change of total body weight .
Grip strength | Baseline and 12 weeks
  Changes of grip strength of both hands measured with a grip dynamometer
Protein metabolic markers | Baseline and 12 weeks
  Changes of protein metabolic makers
Changes in intramuscular fat deposition | Baseline and 12 weeks
  Changes of mean muscle attenuation (MA) at the level of L3 in CT

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, doctor, Study Chair — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan HL, Jia J. Chronic hepatitis B in Asia-new insights from the past decade. J Gastroenterol Hepatol. 2011 Jan;26 Suppl 1:131-7. doi: 10.1111/j.1440-1746.2010.06544.x. PMID 21199524
- [Background] Holecek M. Beta-hydroxy-beta-methylbutyrate supplementation and skeletal muscle in healthy and muscle-wasting conditions. J Cachexia Sarcopenia Muscle. 2017 Aug;8(4):529-541. doi: 10.1002/jcsm.12208. Epub 2017 May 10. PMID 28493406
- [Background] Sinclair M, Gow PJ, Grossmann M, Angus PW. Review article: sarcopenia in cirrhosis--aetiology, implications and potential therapeutic interventions. Aliment Pharmacol Ther. 2016 Apr;43(7):765-77. doi: 10.1111/apt.13549. Epub 2016 Feb 5. PMID 26847265
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Tsien C, Davuluri G, Singh D, Allawy A, Ten Have GA, Thapaliya S, Schulze JM, Barnes D, McCullough AJ, Engelen MP, Deutz NE, Dasarathy S. Metabolic and molecular responses to leucine-enriched branched chain amino acid supplementation in the skeletal muscle of alcoholic cirrhosis. Hepatology. 2015 Jun;61(6):2018-29. doi: 10.1002/hep.27717. Epub 2015 Feb 27. PMID 25613922
- [Background] Wilkinson DJ, Hossain T, Limb MC, Phillips BE, Lund J, Williams JP, Brook MS, Cegielski J, Philp A, Ashcroft S, Rathmacher JA, Szewczyk NJ, Smith K, Atherton PJ. Impact of the calcium form of beta-hydroxy-beta-methylbutyrate upon human skeletal muscle protein metabolism. Clin Nutr. 2018 Dec;37(6 Pt A):2068-2075. doi: 10.1016/j.clnu.2017.09.024. Epub 2017 Oct 6. PMID 29097038
- [Background] Tsien CD, McCullough AJ, Dasarathy S. Late evening snack: exploiting a period of anabolic opportunity in cirrhosis. J Gastroenterol Hepatol. 2012 Mar;27(3):430-41. doi: 10.1111/j.1440-1746.2011.06951.x. PMID 22004479
- [Background] Takaguchi K, Moriwaki H, Doyama H, Iida M, Yagura M, Shimada N, Kang M, Yamada H, Kumada H. Effects of branched-chain amino acid granules on serum albumin level and prognosis are dependent on treatment adherence in patients with liver cirrhosis. Hepatol Res. 2013 May;43(5):459-66. doi: 10.1111/j.1872-034X.2012.01097.x. Epub 2012 Oct 10. PMID 23046471
- [Background] Plank LD, Gane EJ, Peng S, Muthu C, Mathur S, Gillanders L, McIlroy K, Donaghy AJ, McCall JL. Nocturnal nutritional supplementation improves total body protein status of patients with liver cirrhosis: a randomized 12-month trial. Hepatology. 2008 Aug;48(2):557-66. doi: 10.1002/hep.22367. PMID 18627001
- [Background] Nishikawa H, Shiraki M, Hiramatsu A, Moriya K, Hino K, Nishiguchi S. Japan Society of Hepatology guidelines for sarcopenia in liver disease (1st edition): Recommendation from the working group for creation of sarcopenia assessment criteria. Hepatol Res. 2016 Sep;46(10):951-63. doi: 10.1111/hepr.12774. PMID 27481650